CLINICAL TRIAL: NCT01789658
Title: A Randomized Controlled Trial of Cryotherapy for Prevention and Reduction of Severity of Oral Mucositis in Children Undergoing Hematopoietic Stem Cell Transplantation.
Brief Title: Cryotherapy for Prevention of Oral Mucositis in Children Undergoing Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: The Swedish Childhood Cancer Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UU-OM-01
Record Dates: First submitted 2013-02-05; First posted 2013-02-12 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Oral Mucositis; Pain; Infection; Nutrition Aspect of Cancer
Keywords: Oral Mucositis; Children; Cryotherapy; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Stomatitis; Pain; Infections | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cryotherapy (Experimental): Cryotherapy during conditioning treatment with chemotherapy prior to HSCT
  Interventions: Other: Cryotherapy
- Control (No Intervention): Standard oral Care. No Cryotherapy during conditioning treatment prior to HSCT

INTERVENTIONS:
Other: Cryotherapy — Cryotherapy with ice-chips, ice cream or ice water is given during conditioning treatment with chemotherapy prior to HSCT.
  Arms: Cryotherapy

SUMMARY:
Oral mucositis (OM) is a common adverse effect of chemotherapy, radiotherapy and conditioning regimens before Hematopoietic Stem Cell Transplantation (HSCT). The aim of this study is to effectiveness of cryotherapy as a prophylactic treatment in children undergoing HSCT.

DETAILED DESCRIPTION:
There is a complex pathobiology behind OM; chemo and radiotherapy affects the mucosa and submucosa causing DNA-strand brakes and generation of reactive oxygen species (ROS). This initiates a cascade of events, among others activation of transcription factors, up-regulation of pro-inflammatory cytokines, and activation of macrophages and proteases leading to tissue injury causing symptoms such as erythema, edema, ulceration, taste perception alterations, and mouth dryness. OM often causes local and systemic infections, fatigue, pain, and difficulties in basal functions such as swallowing (and hence drinking and eating) and talking and reduces patients' psychological well-being. Nearly 90 % of pediatric patients undergoing HSCT are afflicted with OM. In pediatric patients mucositis is reported as one of the most painful and debilitating side effects during cancer treatment.Beyond a significant suffering for the patient it is hence associated with higher costs for health care and increased mortality.

The current scientific situation regarding prevention and treatment of OM has been summarized in Cochrane reports showing limited data on adults and practically missing data on children and adolescents. Concluding guidelines from these reports emphasize the need for well conducted randomized controlled trials (RCT's) to evaluate and refine treatments in order to establish evidence based interventions.

The use of cryotherapy to prevent oral mucositis in patients who are receiving high-dose chemotherapy as a conditioning agent prior to HSCT continue to show evidence in the adult population.

The aim of this study is to compare treatment with cryotherapy (Arm 1)with a standard oral care protocal (Arm 2)

ARM 1 Children are instructed to use chew on ice-chips, ingest ice-cream or ice-water during infusion of chemotherapy as part of the conditioning treatment prior to HSCT. Melted ice should be replaced by new as soon as possible. Children receiving a 24-hour infusion are instructed to use cryotherapy for one hour 4 times a day.

ARM 2 Standard care for prevention and management of oral mucositis

Primary outcome

* Degree and duration of Oral mucositis

Secondary outcomes

* Oral pain
* Opioid use
* Duration of parenteral nutrition
* Weight loss
* Duration of neutropenic fever
* Duration of antibiotic treatment
* Duration of hospitalization
* Emotional and psychological status
* C reactive protein (CRP) and s-albumin correlation to grade of Oral Mucositis

ELIGIBILITY:
Inclusion Criteria:

Age between 4-18 Undergoing Hematopoietic Stem Cell Transplantation in Sweden sufficient knowledge in swedish to understand the protocols -

Exclusion Criteria:

-

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Mucositis grade - WHO Oral Toxicity Scale | Daily until engraftment, an expected average of 20 days.
  WHO-Oral toxicity scale Grade 0 - No mucositis Grade 1 - Erythema and/or soreness Grade 2 - Erythema and/or ulcers. Can eat solid food. Grade 3 - Erythema and/or Ulcers. No solid food but can ingest liquids. Grade 4 - Oral alimentation not possible.

SECONDARY OUTCOMES:
Mucositis grade - Children´s International Mucositis Evaluation Scale (ChiMES) | Daily until engraftment, an expected average of 20 days.
  Daily evaluation by child and parent.
Pain - Childrens Hospital Eastern Ontario Pain Scale (CHEOPS) | Daily until Engraftment an expected average of 20 days.
  Daily assessment by nurse
Mouth Pain | Daily until Engraftment an expected average of 20 days
  Mouth Pain measured with Numerical Rating scale(NRS)for children >7 years and parents and Facial Pain Scale(FPS) for children < 7 years
Emotional and Psychological status | Daily until engraftment, an expected average of 20 days.
  Beck youth inventories for depression and anxiety

OTHER OUTCOMES:
Opioid consumption | During hospitalization in connection with HSCT, an expected average of 25 days
  Days with, and dose of morphine-equivalent opioids
Duration of parenteral nutrition | During hospitalization in connection with HSCT, an expected average of 25 days
  Days with Total Parenteral Nutrition
Weight Loss | During hospitalization in connection with HSCT, an expected average of 25 days
  Weight Loss in kilograms from admission to date of engraftment
Duration of Antibiotic treatment | During hospitalization in connection with HSCT, an expected average of 25 days
  Days with antibiotics
Duration of febrile neutropenia | Until engraftment, an expected average of 20 days
  Days with fever >38.0 degrees
Duration of Hospitalisation | During hospitalization in connection with HSCT, an expected average of 25 days
  Counted from day 0 until discharge either home or to region hospital.
C reactive protein | During hospitalization in connection with HSCT, an expected average of 25 days
  Level of p-CRP in comparison to grade of mucositis
S-Albumin | During hospitalization in connection with HSCT, an expected average of 25 days
  In correlation to grade of Oral Mucositis

CONTACTS AND LOCATIONS:
Overall Officials: Gustaf Ljungman, MD, PhD, Study Director — Uppsala University
Locations (5):
- Sweden (5):
  - Pediatric Oncology Department, Queen Silvia Childrens´ Hospital, Gothenburg
  - Departent of Pediatric Oncology, Lund University Hospital, Lund
  - Center for Allogeneic Stem Cell Transplantation, Karolinska University Hospital, Hudding, Stockholm
  - Department of pediatrics B78, Karolinska University Hospital, Stockholm
  - Department of Hematology, Uppsala University Hospital, Uppsala

REFERENCES:
- [Derived] Kamsvag T, Svanberg A, Legert KG, Arvidson J, von Essen L, Mellgren K, Toporski J, Winiarski J, Ljungman G. Prevention of oral mucositis with cryotherapy in children undergoing hematopoietic stem cell transplantations-a feasibility study and randomized controlled trial. Support Care Cancer. 2020 Oct;28(10):4869-4879. doi: 10.1007/s00520-019-05258-2. Epub 2020 Jan 28. PMID 31993753